CLINICAL TRIAL: NCT06216652
Title: Enhancing Balance, Strength, Flexibility and Spatiotemporal Gait Parameters in Pediatric Cerebral Palsy: Treadmill Training at Variable Inclinations
Brief Title: Treadmill Training at Variable Inclinations in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Berna Ramanli, assistant professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PamukkaleU-SBF-BR-01
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- downhill walking (Active Comparator): All participants received a conventional physiotherapy program. In addition to this program, the first group performed downhill walking exercise on the treadmill
  Interventions: Other: downhill walking
- uphill walking (Active Comparator): All participants received a conventional physiotherapy program. In addition to this program, the second group performed uphill walking exercise on the treadmill
  Interventions: Other: uphill walking
- walking with no incline (Active Comparator): All participants received a conventional physiotherapy program. In addition to this program, the third group performed walking with no incline exercise on the treadmill
  Interventions: Other: walking with no incline

INTERVENTIONS:
Other: downhill walking — All participants received a conventional physiotherapy program for 2 days/week, 40 min/day for 8 weeks. In addition to this program, the first group performed downhill walking exercise on the treadmill for 2 days/week, 30 min/day on different days.
  Arms: downhill walking
Other: uphill walking — All participants received a conventional physiotherapy program for 2 days/week, 40 min/day for 8 weeks. In addition to this program, the second group performed uphill walking exercise on the treadmill for 2 days/week, 30 min/day on different days.
  Arms: uphill walking
Other: walking with no incline — All participants received a conventional physiotherapy program for 2 days/week, 40 min/day for 8 weeks. In addition to this program, the third group performed walking with no incline walking exercise on the treadmill for 2 days/week, 30 min/day on different days.
  Arms: walking with no incline

SUMMARY:
This study aimed to evaluate the effect of treadmill training (TT) at different inclinations on balance, strength, flexibility, and gait parameters in children with cerebral palsy (CP) in addition to traditional physiotherapy applications.

Forty-two participants with CP aged 7-18 years and at Gross Motor Function Classification System level 2 were randomized into three groups: downhill walking (DW), uphill walking (UW), and walking with no incline (WWI). Balance, isometric strength, flexibility, and gait parameters were assessed at baseline (2nd week) and at 11th week. The groups were provided with TT and conventional treatment.

All groups showed improvement in balance. Isometric strength values showed improvement in knee flexion (KF) on the affected side (AS) in DW and UW groups, and in knee extension force in UW and WWI groups. In flexibility, hip flexion, hip extension and ankle dorsiflexion improved in all groups, while KF and ankle plantar flexion improved only in DW and WWI. Duration of the modified timed up-and-go test showed significant improvements in the DW and UW groups.

TT performed at different inclinations improved balance, isometric strength, flexibility, and gait parameters on both the AS and the nonaffected side.

DETAILED DESCRIPTION:
TT is a therapeutic technique in the rehabilitation of children with CP. Positive effects of different TT protocols have been observed in patients with CP; however, there is no study examining the effects of forward downhill TT. Therefore, this study aimed to investigate the effect of TT with forward downhill walking (DW), forward uphill walking (UW), and forward walking with no incline (WWI) on balance, strength, flexibility, and gait parameters in 7-18-year-old children with hemiparetic and diparetic CP in addition to traditional physiotherapy applications.

Sixty-four participants were initially recruited in this study. However, 42 participants (18 female, 24 male) with hemiparetic and diparetic CP completed the study. The study was conducted in a Special Education and Rehabilitation Center in Denizli, Turkey between April 2021 and June 2022. The inclusion criteria for the study were (a) age between 7-18 yrs old, (b) being at Gross Motor Functional Classification System (GMFCS) levels II, (c) no cooperation problems that would interfere with communication, (d) no surgical treatment or neuromuscular injection in the last 6 months (e) no unstoppable epileptic seizures, (f) asymmetric lower extremity shortness >4 cm and no any health problems except CP. Exclusion criteria from the study were trauma during the study period, not participating in the exercise program by more than 20%, willing to quit voluntarily, having a spasticity ≥2 on the Modified Ashworth Scale (MAS) measured from the lower extremity All parents/guardians agreed to the participation of their children by signing a statement of informed consent. The investigation was approved by the Pamukkale University Clinical Research Ethics Committee (60116787-020-35801/24.03.2021). All procedures were realized in according to the Declaration of Helsinki.

To ensure that the gender and age distributions to be observed in the groups were similar, a randomization table was prepared by stratified randomization method before the study.

All participants received a conventional physiotherapy program for 2 days/week, 40 min/day for 8 weeks. In addition to this program, the first group performed DW TT, the second group performed UW TT, and the third group performed WWI TT walking exercise on the treadmill for 2 days/week, 30 min/day on different days. At the beginning and end of the 8-week program, the participants' lower extremity isometric strength was assessed using a hand-held dynamometer, dynamic balance was assessed using a functional reach test (FRT), flexibility was assessed range of motion (ROM) using a goniometer, and gait performance was assessed using a spatiotemporal gait analyzer. All measurements included familiarization trials. Conventional physiotherapy program, walking exercises, and measurements were conducted in standard conditions (22-25 °C, 25%-45% relative humidity) during the morning hours in a quiet room by the same physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* age between 7-18 yrs old,
* being at Gross Motor Functional Classification System (GMFCS) levels II,
* no cooperation problems that would interfere with communication,
* no surgical treatment or neuromuscular injection in the last 6 months
* no unstoppable epileptic seizures,
* asymmetric lower extremity shortness >4 cm and no any health problems except CP.

Exclusion criteria:

* trauma during the study period,
* not participating in the exercise program by more than 20%, willing to quit voluntarily,
* having a spasticity ≥2 on the Modified Ashworth Scale (MAS) measured from the lower extremity

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Dynamic balance was assessed using the functional reach test (FRT), one of the physical fitness parameters, which is a reliable and valid assessment tool for assessing balancing ability among children with CP. The results were recorded in centimeters and statistics were made on their averages.
Isometric muscle strength | 8 weeks
  The isometric muscle strength, one of the physical fitness parameters, is a reliable assessment tool for assessing isometric strength among children with CP. The isometric muscle strength of the participants' knee flexor and extensor muscles was evaluated with a hand dynamometer (JTECH Medical PowerTrack II Commander, Salt Lake City, UT, USA). The results were recorded in newton and statistics were made on their averages.
Flexibility | 8 weeks
  Range of motion measurements, one of the physical fitness parameters, were performed manually with a goniometer. The results were recorded in degree and statistics were made on their averages.
Spatiotemporal gait analysis | 8 weeks
  Gait performance, one of the physical fitness parameters, was assessed with the LEGSystm spatiotemporal gait analyzer (LegSys/BioSenics, Watertown, USA). The results were recorded as time (s and min), distance (m) and step frequency (step/min), and statistics were made on their averages.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Ramanlı, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)